CLINICAL TRIAL: NCT01113801
Title: A Randomized, Double-Masked, Placebo-Controlled, Multicenter, Phase 2 Study to Evaluate the Safety and Renal Efficacy of LY2382770 in Patients With Diabetic Kidney Disease Due to Type 1 or Type 2 Diabetes
Brief Title: A Study in Participants With Diabetic Kidney Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Interim Assessment: Lack of Efficacy
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 10168; H9V-MC-GFRF (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-04-28; First posted 2010-04-30 (Estimated); Results first posted 2017-12-13 (Actual); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Diabetic Kidney Disease; Diabetic Nephropathy; Diabetic Glomerulosclerosis
Keywords: Chronic Kidney Disease; Diabetic Kidney Disease; End-Stage Renal Disease; Transforming Growth Factor beta 1 Monoclonal Antibody; Type 1 Diabetes; Type 2 Diabetes
MeSH Terms: conditions — Diabetic Nephropathies; Renal Insufficiency, Chronic; Kidney Failure, Chronic; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- 2 mg LY2382770 (Experimental)
  Interventions: Drug: LY2382770
- 10 mg LY2382770 (Experimental)
  Interventions: Drug: LY2382770
- 50 mg LY2382770 (Experimental)
  Interventions: Drug: LY2382770

INTERVENTIONS:
Drug: LY2382770 — Subcutaneous injection given monthly for 12 months
  Arms: 10 mg LY2382770; 2 mg LY2382770; 50 mg LY2382770
Drug: Placebo — Subcutaneous injection given monthly for 12 months
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if LY2382770 is safe and effective at protecting kidney function in participants with kidney disease due to diabetes.

DETAILED DESCRIPTION:
The primary objective is to determine if LY2382770, administered monthly for 1 year, is more effective than placebo at slowing the progression of diabetic kidney disease in participants treated with an angiotensin-converting enzyme inhibitor (ACEi) or an angiotensin II receptor blocker (ARB).

ELIGIBILITY:
Main Inclusion Criteria:

* Participants with chronic kidney disease presumed due to diabetes Type 1 or Type 2
* Participants with certain levels of kidney function - serum creatinine (SCr) 1.3 to 3.3 mg/dl (115 to 291 micromol/L) inclusive for women and 1.5 to 3.5 mg/dl (132 to 309 micromol/L) inclusive for men, or an estimated glomerular filtration rate (eGFR) 20 to 60 mL/min/1.73 m²
* Participants with protein in the urine - 24-hour urine protein/creatinine ratio (PCR) greater than or equal to 800 mg/g (greater than or equal to 91 mg/mmol).
* Participants must be on a stable and acceptable dose of an ACE (angiotensin-converting enzyme) inhibitor or an ARB (angiotensin II receptor blocker), or not able to tolerate these medications.

Main Exclusion Criteria:

* Female participants who can become pregnant, are pregnant or breastfeeding
* Participants who have any of the following medical conditions (the site research staff will discuss these criteria and determine a participant's ability to participate)

  * Chronic inflammatory or autoimmune diseases
  * Chronic Kidney Disease from causes other than diabetes
  * An organ transplant
  * Too high a blood pressure
  * Viral Hepatitis B or C liver infection, liver cirrhosis, or significant liver disease
  * Recent gastrointestinal bleeding
  * Acute kidney injury within the 3 months before screening
  * Major surgery within 3 months before screening or plan to have it during the study period
  * HIV infection- the virus that causes AIDS
  * Heart disease that is not considered stable
  * Cancer that is too recent or other condition which poses too high a risk for developing cancer
  * Required to take drugs that change the immune system

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 417 (Actual)
Dates: Start 2010-07; Primary Completion 2014-05 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (78):
- United States (28):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Phoenix, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Inglewood, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Los Angeles, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Northridge, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Denver, Colorado
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Port Charlotte, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tampa, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Atlanta, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Idaho Falls, Idaho
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wichita, Kansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kenner, Louisiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rockville, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kansas City, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Omaha, Nebraska
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chapel Hill, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Charlotte, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Durham, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Greenville, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Winston-Salem, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Beachwood, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bend, Oregon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Providence, Rhode Island
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Orangeburg, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dallas, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lufkin, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., St. George, Utah
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Suffolk, Virginia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Milwaukee, Wisconsin
- Australia (13):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Camperdown, New South Wales
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Concord, New South Wales
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gosford, New South Wales
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Liverpool, New South Wales
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Adelaide, South Australia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Launceston, Tasmania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Box Hill, Victoria
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fitzroy, Victoria
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Heidelberg, Victoria
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Melbourne, Victoria
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Parkville, Victoria
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Reservoir, Victoria
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nedlands, Western Australia
- Czechia (8):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Český Krumlov
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Děčín
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jilemnice
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Liberec
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ostrava
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Prague
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tábor
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Teplice
- France (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Grenoble
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lyon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nanterre
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Valenciennes
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vandœuvre-lès-Nancy
- Hungary (10):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Baja
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Balatonfüred
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Budapest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gyöngyös
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Győr
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kaposvár
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nagykanizsa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Szeged
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Szigetvár
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Zalaegerszeg
- Israel (12):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ashkelon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hadera
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Haifa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Holon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jerusalem
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kfar Saba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nahariya
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rehovot
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Safed
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tel Aviv
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tel Litwinsky
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ẕerifin
- Puerto Rico (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cidra
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rio Piedras

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo given subcutaneous (SC) injection monthly for 12 months
- 2 mg LY2382770: 2 milligrams (mg) LY2382770 given (SC) injection monthly for 12 months
- 10 mg LY2382770: 10 mg LY2382770 given SC injection monthly for 12 months
- 50 mg LY2382770: 50 mg LY2382770 given SC injection monthly for 12 months
Period: Overall Study
Arm/Group | Placebo | 2 mg LY2382770 | 10 mg LY2382770 | 50 mg LY2382770
Started | 103 | 105 | 103 | 106
Received at Least One Dose of Drug | 103 | 105 | 103 | 105
Completed | 62 | 65 | 66 | 65
Not Completed | 41 | 40 | 37 | 41
Not completed — Adverse Event | 4 | 0 | 2 | 6
Not completed — Death | 4 | 5 | 3 | 4
Not completed — Protocol Violation | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 9 | 7 | 7 | 8
Not completed — Physician Decision | 2 | 2 | 3 | 3
Not completed — Sponsor Decision | 15 | 21 | 20 | 15
Not completed — Clinical Endpoint (ESRD) | 7 | 4 | 2 | 5

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 2 mg LY2382770 | 10 mg LY2382770 | 50 mg LY2382770 | Total
Number analyzed (Participants) | 103 | 105 | 103 | 105 | 416
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.7 (11.31) | 62.8 (9.20) | 60.5 (9.05) | 62.9 (10.86) | 62.2 (10.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 21 | 29 | 19 | 96
  Male | 76 | 84 | 74 | 86 | 320
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 11 | 11 | 15 | 45
  Not Hispanic or Latino | 55 | 58 | 53 | 45 | 211
  Unknown or Not Reported | 40 | 36 | 39 | 45 | 160
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 4 | 2 | 2 | 8
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1 | 0 | 2
  Black or African American | 14 | 9 | 9 | 7 | 39
  White | 83 | 90 | 84 | 90 | 347
  More than one race | 1 | 0 | 2 | 0 | 3
  Unknown or Not Reported | 4 | 2 | 5 | 6 | 17
Region of Enrollment [Count of Participants; unit: Participants]
  France | 8 | 9 | 7 | 8 | 32
  United States | 37 | 35 | 38 | 36 | 146
  Czechia | 14 | 9 | 10 | 12 | 45
  Hungary | 11 | 16 | 15 | 15 | 57
  Puerto Rico | 3 | 5 | 2 | 5 | 15
  Australia | 10 | 10 | 10 | 10 | 40
  Israel | 20 | 21 | 21 | 20 | 82
Serum Creatinine [Mean (Standard Deviation); unit: milligram/deciliter (mg/dl)] | 2.209 (0.5917) | 2.127 (0.5824) | 2.091 (0.6538) | 2.132 (0.6289) | 2.140 (0.6141)
Urine Protein/Creatinine Ratio [Mean (Standard Deviation); unit: gram/gram] | 3.123 (2.5180) | 3.266 (2.5723) | 3.301 (2.4510) | 3.354 (2.5457) | 3.262 (2.5148)
Estimated Glomerular Filtration Rate (eGFR) [Mean (Standard Deviation); unit: milliliter/minute/1.73 meter squared] | 33.835 (11.0568) | 35.705 (11.7226) | 36.358 (12.5154) | 35.945 (12.0852) | 35.464 (11.8539)

OUTCOME MEASURES:

1. Primary Outcome: Change in Log Transformed (In) Serum Creatinine From Baseline to 12 Month Endpoint
Description: Analysis of covariance (ANCOVA) model was used with treatment, visit, and treatment-by-visit interaction as fixed effects, subject as random effect, baseline Serum Creatinine log transformed (ln) and first morning urine protein to creatinine ratio (PCR) log transformed (ln) as covariates.
Time Frame: Baseline, 12 months
Population: All randomized participants who received at least 1 dose of drug and had evaluable baseline and post baseline serum creatinine values.
Measure: Least Squares Mean (Standard Error); unit: ln milligrams per deciliter [ln(mg/dL)]
Groups:
- 2 mg LY2382770: 2 mg LY2382770 given (SC) injection monthly for 12 months
Arm/Group | Placebo | 2 mg LY2382770 | 10 mg LY2382770 | 50 mg LY2382770
Number analyzed (Participants) | 85 | 90 | 91 | 82
ln milligrams per deciliter [ln(mg/dL)] | 0.13 (0.019) | 0.18 (0.019) | 0.17 (0.019) | 0.17 (0.020)

2. Secondary Outcome: Change in Log Transformed (ln) Urine Protein/Creatinine Ratio From Baseline to 12 Month Endpoint
Description: as for outcome 1
Time Frame: Baseline, 12 months
Population: All randomized participants who received at least 1 dose of drug and had evaluable urine protein and creatinine ratio values.
Measure: Least Squares Mean (Standard Error); unit: ln grams/grams [ln( g/g)]
Arm/Group | Placebo | 2 mg LY2382770 | 10 mg LY2382770 | 50 mg LY2382770
Number analyzed (Participants) | 82 | 87 | 85 | 81
ln grams/grams [ln( g/g)] | 0.06 (0.076) | 0.05 (0.072) | 0.05 (0.073) | -0.01 (0.075)

3. Secondary Outcome: Population Pharmacokinetics (PK) - Model-Estimated Area Under the Concentration -Time Curve (AUC ) Over a Dosing Interval
Time Frame: Baseline through 12 months (samples collected pre and/or postdose at monthly intervals)
Population: All randomized participants who received at least 1 dose of drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram*hour per milliliter(µg•hr/mL)
Arm/Group | Placebo | 2 mg LY2382770 | 10 mg LY2382770 | 50 mg LY2382770
Number analyzed (Participants) | 0 | 105 | 101 | 104
microgram*hour per milliliter(µg•hr/mL) |  | 54.4 (49) | 197 (45) | 957 (44)

4. Secondary Outcome: Log Transformed (ln) Serum Creatinine Slope of Change From Baseline Through 12 Months
Description: Analysis of covariance (ANCOVA) model was used with treatment as fixed effects and baseline Serum Creatinine log transformed (ln) and first morning urine protein to creatinine ratio (PCR) log transformed (ln) as covariates.
Time Frame: Baseline through 12 months
Population: All randomized participants who received at least 1 dose of drug.
Measure: Least Squares Mean (Standard Error); unit: ln milligrams per deciliter(mg/dL)/month
Arm/Group | Placebo | 2 mg LY2382770 | 10 mg LY2382770 | 50 mg LY2382770
Number analyzed (Participants) | 103 | 105 | 103 | 105
ln milligrams per deciliter(mg/dL)/month | 0.01605 (0.002685) | 0.01408 (0.002731) | 0.01716 (0.002658) | 0.01337 (0.002712)

5. Secondary Outcome: Estimated Glomerular Filtration Rate (eGFR) Slope of Change From Baseline Through 12 Months
Description: Analysis of covariance (ANCOVA) model was used with treatment as fixed effects, baseline Serum Creatinine log transformed (ln) and first morning urine protein to creatinine ratio (PCR) ) log transformed (ln) as covariates.
Time Frame: Baseline through 12 months
Population: All randomized participants who received at least 1 dose of drug.
Measure: Least Squares Mean (Standard Error); unit: mL/min/1.73 m²/month
Arm/Group | Placebo | 2 mg LY2382770 | 10 mg LY2382770 | 50 mg LY2382770
Number analyzed (Participants) | 103 | 105 | 103 | 105
mL/min/1.73 m²/month | -0.3727 (0.08599) | -0.3664 (0.08742) | -0.5554 (0.08512) | -0.3980 (0.08683)

ADVERSE EVENTS:
Description: All randomized participants who received at least 1 dose of drug. All serious adverse events following randomization are reported.
Arm/Group | Placebo | 2 mg LY2382770 | 10 mg LY2382770 | 50 mg LY2382770
Serious Adverse Events (participants affected / at risk) | 39/103 | 44/105 | 37/103 | 41/105
Other Adverse Events (participants affected / at risk) | 57/103 | 67/105 | 62/103 | 62/105
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo (N=103) | 2 mg LY2382770 (N=105) | 10 mg LY2382770 (N=103) | 50 mg LY2382770 (N=105)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 1 (1) | 2 (2)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Acute myocardial infarction (Cardiac disorders) | 3 (3) | 4 (5) | 1 (1) | 3 (5)
Angina pectoris (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Angina unstable (Cardiac disorders) | 0 (0) | 2 (3) | 2 (2) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 5 (5) | 1 (1) | 3 (3) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 2 (2) | 0 (0) | 4 (4) | 6 (8)
Cardiomegaly (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Mitral valve disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 2 (2) | 2 (2) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Corneal oedema (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Macular hole (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Posterior capsule rupture (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Retinal artery occlusion (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vitreous haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (4)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Gastrointestinal inflammation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Inguinal hernia, obstructive (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intestinal polyp (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mallory-weiss syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Device failure (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Generalised oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Multi-organ failure (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sudden death (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Liver disorder (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Breast abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchiolitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchopneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 2 (4) | 2 (2) | 2 (2) | 2 (3)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dermatitis infected (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Enterobacter bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Furuncle (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gangrene (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Infective exacerbation of bronchiectasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intervertebral discitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Klebsiella sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Orchitis (Infections and infestations) | 0/76 (0) | 1/84 (1) | 0/74 (0) | 0/86 (0)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Otitis externa (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 4 (4)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia staphylococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pseudomembranous colitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Staphylococcal abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Streptococcal urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Superinfection bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arteriovenous fistula occlusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Postoperative thoracic procedure complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary retention postoperative (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 1 (1) | 1 (3) | 1 (1) | 1 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (2) | 2 (2) | 0 (0) | 1 (1)
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 1 (1) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (3) | 1 (1) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myopathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neuropathic arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sweat gland tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Central nervous system lesion (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebellar ischaemia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 3 (3) | 1 (1) | 1 (1)
Diabetic hyperosmolar coma (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diabetic mononeuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hemiparesis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hydrocephalus (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemic coma (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemic seizure (Nervous system disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Ischaemic cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Vertebrobasilar insufficiency (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Azotaemia (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetic nephropathy (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nephropathy (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 2 (2) | 1 (1) | 2 (2)
Renal failure acute (Renal and urinary disorders) | 2 (3) | 5 (5) | 3 (3) | 8 (10)
Renal failure chronic (Renal and urinary disorders) | 5 (5) | 4 (4) | 2 (2) | 1 (1)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Arteriosclerosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vena cava thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo (N=103) | 2 mg LY2382770 (N=105) | 10 mg LY2382770 (N=103) | 50 mg LY2382770 (N=105)
Anaemia (Blood and lymphatic system disorders) | 7 (7) | 6 (6) | 4 (4) | 5 (5)
Constipation (Gastrointestinal disorders) | 4 (4) | 8 (10) | 8 (8) | 5 (7)
Diarrhoea (Gastrointestinal disorders) | 4 (8) | 10 (15) | 11 (14) | 6 (6)
Nausea (Gastrointestinal disorders) | 5 (5) | 7 (8) | 5 (5) | 7 (8)
Vomiting (Gastrointestinal disorders) | 4 (4) | 3 (3) | 5 (6) | 8 (10)
Fatigue (General disorders) | 8 (9) | 3 (3) | 6 (6) | 5 (5)
Local swelling (General disorders) | 7 (7) | 2 (3) | 1 (2) | 1 (2)
Oedema peripheral (General disorders) | 15 (15) | 20 (22) | 11 (11) | 5 (5)
Bronchitis (Infections and infestations) | 5 (5) | 8 (8) | 4 (4) | 6 (6)
Influenza (Infections and infestations) | 4 (4) | 6 (8) | 4 (4) | 2 (2)
Nasopharyngitis (Infections and infestations) | 8 (8) | 6 (6) | 3 (5) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 10 (11) | 11 (11) | 13 (16) | 11 (13)
Urinary tract infection (Infections and infestations) | 6 (6) | 10 (11) | 1 (2) | 3 (3)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 6 (6) | 8 (8) | 4 (4)
Hypoglycaemia (Metabolism and nutrition disorders) | 10 (16) | 13 (20) | 9 (25) | 7 (15)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (5) | 7 (8) | 6 (7) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 8 (8) | 9 (9) | 5 (5)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 (3) | 6 (6) | 4 (5) | 4 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4) | 8 (11) | 4 (4) | 5 (6)
Dizziness (Nervous system disorders) | 8 (9) | 8 (9) | 4 (4) | 9 (12)
Headache (Nervous system disorders) | 3 (5) | 7 (7) | 8 (9) | 2 (2)
Uterine polyp (Reproductive system and breast disorders) | 0/27 (0) | 0/21 (0) | 0/29 (0) | 1/19 (1)
Vaginal discharge (Reproductive system and breast disorders) | 0/27 (0) | 0/21 (0) | 0/29 (0) | 1/19 (1)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0/27 (0) | 0/21 (0) | 0/29 (0) | 1/19 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 7 (7) | 5 (6) | 9 (10)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (4) | 2 (2) | 6 (6)
Hypertension (Vascular disorders) | 6 (6) | 6 (6) | 9 (9) | 5 (5)

LIMITATIONS AND CAVEATS:
Study was stopped early for efficacy futility per recommendation by the independent Data Safety Monitoring Committee.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days